CLINICAL TRIAL: NCT05925790
Title: Observational Study on Anti-interleukin-1 Receptor Antagonist Antibodies and Soluble Urokinase Plasminogen Activator Receptor (suPAR) in Pericarditis: PERIPLO (PERicarditis: IL-1 RA Antibodies and suPAR Levels Observational) Study
Brief Title: Clinical Phenotypes in Pericarditis: IL-1RA Antibodies and suPAR Levels
Acronym: PERIPLO
Status: Recruiting | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Fatebenefratelli Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale Galeazzi Sant'Ambrogio - IRCCS (Unknown); Careggi Hospital (Other); Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other); Children's Medical Hospital, University of Muenster, Muenster, Germany (Other); University of Homburg (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Maddalena Alessandra Wu, MD, ASST Fatebenefratelli Sacco
Other Study IDs: 2023/ST/094
Record Dates: First submitted 2023-05-28; First posted 2023-06-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pericarditis
Keywords: Pericarditis; Anti-interleukin-1 receptor antagonist antibodies; Soluble urokinase plasminogen activator receptor; Pericarditis phenotypes
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be withdrawn to test:
  * IL-1RA Antibodies;
  * suPAR levels;
  * biochemical tests used in routine clinical practice, including complete blood count, biochemistry panel (C-reactive protein, urea, creatinine, sodium, potassium, chloride, calcium, magnesium, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, gamma-glutamyl transferase (gamma-GT), lactate dehydrogenase (LDH), creatine phosphokinase (CPK), albumin, serum iron, transferrin, ferritin, triglycerides, cholesterol + HDL), and coagulation parameters (prothrombin time - PT, activated partial thromboplastin Time - aPTT, fibrinogen, D-dimer).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory phenotype: Patients with the inflammatory phenotype of recurrent pericarditis exhibit signs indicating the presence of an inflammatory process during a recurrence. These signs may include one or more of the following:
  * Fever
  * Elevated C-reactive protein (CRP)
  * Elevated white blood cell (WBC) count
  * Elevated erythrocyte sedimentation rate (ESR)
  * Pericardial late gadolinium enhancement (LGE) on cardiac magnetic resonance imaging (CMR)
  * Pericardial contrast enhancement on computed tomography (CT)
  Interventions: Diagnostic Test: IL1RA Antibody Assay; Diagnostic Test: suPAR Testing
- Non-inflammatory phenotype: Patients with the non-inflammatory phenotype of recurrent pericarditis do not exhibit any of the signs typically associated with an active inflammatory process during a recurrence. These patients present without:
  * Fever
  * Elevated CRP
  * Elevated WBC count
  * Elevated ESR
  * Pericardial LGE on CMR
  * Pericardial contrast enhancement on CT
  Interventions: Diagnostic Test: IL1RA Antibody Assay; Diagnostic Test: suPAR Testing

INTERVENTIONS:
Diagnostic Test: IL1RA Antibody Assay — -The measurement of anti-interleukin-1 receptor antagonist (IL1RA) antibodies will be performed using the ELISA (Enzyme-Linked Immunosorbent Assay) method,as previously described [Thurner, L., et al., IL-1RA Antibodies in Myocarditis after SARS-CoV-2 Vaccination. N Engl J Med, 2022. 387(16): p. 1524-1527].
Diagnostic Test: suPAR Testing — -The quantitative determination of soluble urokinase plasminogen activator receptor (suPAR) levels in blood will be conducted using the commercially available "CHORUS suPAR Extended" kit (cod. 81414, DIESSE Diagnostica Senese S.p.A., Siena, Italy), based on the principle of the sandwich ELISA method.

SUMMARY:
This study aims to investigate the pathophysiology of recurrent pericarditis (RP) by testing for neutralizing autoantibodies against interleukin-1 receptor antagonist (IL-1RA) and measuring soluble urokinase plasminogen activator receptor (suPAR) levels. The hypothesis is that these tests will provide insights into both the inflammatory and non-inflammatory phenotypes of RP, shedding light on the underlying mechanisms. The study will assess the correlation between antibody levels, suPAR levels, and markers of cardiac damage and inflammation. Longitudinal testing during acute episodes and intercritical phases is also planned. The results may guide the use of anakinra, an IL-1 receptor antagonist, in specific clinical scenarios and optimize treatment strategies for RP.

DETAILED DESCRIPTION:
Recurrent pericarditis (RP) is a complex challenging condition, which significantly impacts patients' quality of life, both from the physical and emotional point of view, and can lead to dangerous complications such as cardiac tamponade and constrictive pericarditis. Moreover, patients experiencing several recurrences also tend to need substantial healthcare resources without necessarily experiencing clinical improvement. Understanding more into details the pathophysiology underlying RP is certainly of pivotal importance for optimizing workup strategies and treatment protocols. It is now recognized that pericarditis stems from a bidirectional cross-talk between environmental triggers and the innate and adaptive immune systems in a genetically susceptible host, with a central role of the pro-inflammatory agonistic molecule IL-1 (IL-1α and IL-1β) and the so-called inflammasome.

Neutralizing autoantibodies have been identified targeting the endogenous interleukin-1 receptor antagonist (IL-1RA) in conditions characterized by severe systemic inflammation such as myocarditis after Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) vaccination, Coronavirus Disease (COVID-19) and Multisystem Inflammatory Syndrome (MIS-C). Therefore, it is possible to hypothesize that testing patients with RP for these antibodies might add significant insights into the knowledge of the pathophysiology of this condition. This may help uncover different underlying mechanisms with similar clinical presentations. New mechanisms involving hyperphosphorylation of IL-1RA precede peripheral immune tolerance breakdown, which may also contribute to certain pericarditis phenotypes.

Therefore, it is possible to hypothesize that IL-1RA antibody testing could provide important information to better profile RP patients with an inflammatory phenotype (as indicated by common biochemical markers like CRP) and those with a complicated clinical course. These patients often exhibit marked activation of the IL-1 signaling pathway, and IL-1RA antibody testing may help uncover underlying mechanisms and improve their characterization. Given the negative correlation between neutralizing antibodies against IL-1RA (and low circulating levels of IL-1RA) and markers of cardiac damage and inflammation, testing these antibodies in RP might be of value. High titers of IL-1RA antibodies in RP may indicate uncontrolled activation of the IL-1 pathway, shedding light on why some patients experience recurrences when tapering treatment with the naturally occurring IL-1 receptor antagonist, anakinra. Testing these IL-1RA antibodies in other types of pericarditis could also help explore their correlation with clinical phenotypes, including presentation, clinical course, and response to treatment strategies. Key exclusion criteria include pericarditis secondary to specific etiologies (except post-cardiac injury), history of immunosuppression, and any clinical conditions that may influence the results.

Additionally, suPAR testing can complementarily highlight chronic low-grade inflammation, which may underlie certain pericarditis cases that do not exhibit an overt "inflammatory phenotype" (e.g., normal CRP) but are challenging to manage.

Longitudinal testing of patients during acute episodes and intercritical phases is planned if feasible.

In both IL-1RA antibody and suPAR testing, this study aims to provide more accurate markers compared to commonly used markers for the "inflammatory phenotype" and potentially uncover unknown pathophysiological mechanisms. Currently, there is a lack of literature on this topic.

The results of this study may provide a rationale for the selective use of anakinra in specific clinical scenarios and/or guide the evaluation of its dosing with an individualized approach.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patients aged ≥ 18 years before any evaluation is performed.
* Written informed consent from parents or legal guardian and assent from minors aged under 18 years before any evaluation is performed.
* Recurrent acute pericarditis during the acute phase of the disease. The diagnosis of pericarditis is based on the presence of at least two of the following criteria: typical pericarditic chest pain (acute and pleuritic, worsened by positional changes or breathing), pericardial friction rub, diffuse ST segment elevation or PR depressions not previously reported, and pericardial effusion.
* Post-cardiac injury pericarditis (e.g., post-cardiac surgery) that is new or worsening. Recurrence is diagnosed based on the same criteria.

In all patients, the previous history of CRP values should be known to distinguish individuals with inflammatory forms (characterized by significantly elevated CRP values in the clinical history) from those with pericarditis and normal or near-normal CRP levels (clinical history of normal or at most less than 2 times the normal value).

The acute phase of the disease is defined as follows: for pericarditis forms with elevated CRP, the presence of a CRP that is at least double the normal value of the test. For forms with normal CRP, it is based on clinical judgment, as there are no other recognized and validated criteria.

Exclusion Criteria:

* Specific etiologies, including tuberculosis, neoplastic or purulent etiologies, post-cardiac injury syndromes, and autoimmune rheumatic diseases.
* Subjects under 18 years of age.
* Pregnant or lactating women.
* History of immunosuppression, including a positive result on HIV screening tests (ELISA and Western blot).
* Positive QuantiFERON test (QFT-Tuberculosis G In-Tube) or positive Purified Protein Derivative (PPD) test after the initial clinical evaluation.
* History of other significant medical conditions that, according to the investigator, could compromise the outcome or interpretation of the results (e.g., systemic diseases that are not directly the cause of pericarditis but may cause a state of chronic inflammation).
* Use of any medication that the investigator believes could alter the result of the tests to be performed (except those used for the treatment of pericarditis).

Throughout the study, patients will continue to receive the most appropriate therapies for their clinical condition, following current guidelines and good clinical practice, without the participation in the study prejudicing or influencing the choice of therapeutic strategies to be employed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with different phenotypes of pericarditis
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of IL-1RA antibodies across pericarditis phenotypes | 24 months
  * Levels of anti-IL-1RA antibodies in different phenotypes of pericarditis.
  * Levels of anti-IL-1RA antibodies during acute episodes and intercritical phases.
Assessment of suPAR levels across pericarditis phenotypes | 24 months
  * Levels of suPAR in acute and recurrent pericarditis with normal C-reactive protein (CRP).
  * Levels of suPAR during acute episodes and intercritical phases.

SECONDARY OUTCOMES:
Correlation of Time to Recurrence and Disease Activity with Anti-IL-1RA Antibodies in Pericarditis | 24 months
  * Correlate the time to recurrence with the levels of anti-IL-1RA antibodies.
  * Correlate overall disease activity indices with the levels of anti-IL-1RA antibodies.
Correlation of Time to Recurrence and Disease Activity with suPAR Levels in Pericarditis | 24 months
  * Correlate the time to recurrence with the levels of suPAR.
  * Correlate overall disease activity indices with the levels of suPAR.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena A Wu, Principal Investigator — ASST Fatebenefratelli Sacco; Antonio L Brucato, Study Director — Fatebenefratelli Hospital
Locations (9):
- Germany (3):
  - Saarland University, Homburg
  - University Children's Hospital Muenster, Münster
  - University Hospital Tübingen, Tübingen
- Italy (6):
  - A.O.U. Careggi, Florence
  - Luigi Sacco Hospital - ASST Fatebenefratelli Sacco, Milan
  - Fatebenefratelli Hospital - ASST Fatebenefratelli Sacco, Milan
  - Ospedale Galeazzi Sant'Ambrogio - IRCCS, Poliambulatorio Cardiovascolare Cardiologia Universitaria, Milan
  - Policlinico di Milano Ospedale Maggiore, Fondazione IRCCS Ca' Granda, Milan
  - Ospedale Santa Maria della Misericordia dell'ASU-FC, Udine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thurner L, Kessel C, Fadle N, Regitz E, Seidel F, Kindermann I, Lohse S, Kos I, Tschope C, Kheiroddin P, Kiblboeck D, Hoffmann MC, Bette B, Carbon G, Cetin O, Preuss KD, Christofyllakis K, Bittenbring JT, Pickardt T, Fischer Y, Thiele H, Baldus S, Stangl K, Steiner S, Gietzen F, Kerber S, Deneke T, Jellinghaus S, Linke A, Ibrahim K, Grabmaier U, Massberg S, Thilo C, Greulich S, Gawaz M, Mayatepek E, Meyer-Dobkowitz L, Kindermann M, Birk E, Birk M, Lainscak M, Foell D, Lepper PM, Bals R, Krawczyk M, Mevorach D, Hasin T, Keren A, Kabesch M, Abdul-Khaliq H, Smola S, Bewarder M, Thurner B, Bohm M, Pfeifer J, Klingel K. IL-1RA Antibodies in Myocarditis after SARS-CoV-2 Vaccination. N Engl J Med. 2022 Oct 20;387(16):1524-1527. doi: 10.1056/NEJMc2205667. Epub 2022 Sep 21. No abstract available. PMID 36130012
- [Background] Chiabrando JG, Bonaventura A, Vecchie A, Wohlford GF, Mauro AG, Jordan JH, Grizzard JD, Montecucco F, Berrocal DH, Brucato A, Imazio M, Abbate A. Management of Acute and Recurrent Pericarditis: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jan 7;75(1):76-92. doi: 10.1016/j.jacc.2019.11.021. PMID 31918837
- [Background] Lopalco G, Rigante D, Cantarini L, Imazio M, Lopalco A, Emmi G, Venerito V, Fornaro M, Frediani B, Nivuori M, Brucato A, Iannone F. The autoinflammatory side of recurrent pericarditis: Enlightening the pathogenesis for a more rational treatment. Trends Cardiovasc Med. 2021 Jul;31(5):265-274. doi: 10.1016/j.tcm.2020.04.006. Epub 2020 May 3. PMID 32376492
- [Background] Mauro AG, Bonaventura A, Vecchie A, Mezzaroma E, Carbone S, Narayan P, Potere N, Cannata A, Paolini JF, Bussani R, Montecucco F, Sinagra G, Van Tassel BW, Abbate A, Toldo S. The Role of NLRP3 Inflammasome in Pericarditis: Potential for Therapeutic Approaches. JACC Basic Transl Sci. 2021 Feb 22;6(2):137-150. doi: 10.1016/j.jacbts.2020.11.016. eCollection 2021 Feb. PMID 33665514
- [Background] Adler Y, Charron P, Imazio M, Badano L, Baron-Esquivias G, Bogaert J, Brucato A, Gueret P, Klingel K, Lionis C, Maisch B, Mayosi B, Pavie A, Ristic AD, Sabate Tenas M, Seferovic P, Swedberg K, Tomkowski W; ESC Scientific Document Group. 2015 ESC Guidelines for the diagnosis and management of pericardial diseases: The Task Force for the Diagnosis and Management of Pericardial Diseases of the European Society of Cardiology (ESC)Endorsed by: The European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2015 Nov 7;36(42):2921-2964. doi: 10.1093/eurheartj/ehv318. Epub 2015 Aug 29. No abstract available. PMID 26320112
- [Background] Klein A, Cremer P, Kontzias A, Furqan M, Tubman R, Roy M, Lim-Watson MZ, Magestro M. US Database Study of Clinical Burden and Unmet Need in Recurrent Pericarditis. J Am Heart Assoc. 2021 Aug 3;10(15):e018950. doi: 10.1161/JAHA.120.018950. Epub 2021 Jul 21. PMID 34284595
- [Background] Brucato A, Imazio M, Gattorno M, Lazaros G, Maestroni S, Carraro M, Finetti M, Cumetti D, Carobbio A, Ruperto N, Marcolongo R, Lorini M, Rimini A, Valenti A, Erre GL, Sormani MP, Belli R, Gaita F, Martini A. Effect of Anakinra on Recurrent Pericarditis Among Patients With Colchicine Resistance and Corticosteroid Dependence: The AIRTRIP Randomized Clinical Trial. JAMA. 2016 Nov 8;316(18):1906-1912. doi: 10.1001/jama.2016.15826. PMID 27825009
- [Background] Imazio M, Andreis A, De Ferrari GM, Cremer PC, Mardigyan V, Maestroni S, Luis SA, Lopalco G, Emmi G, Lotan D, Marcolongo R, Lazaros G, De Biasio M, Cantarini L, Dagna L, Cercek AC, Pivetta E, Varma B, Berkson L, Tombetti E, Iannone F, Prisco D, Caforio ALP, Vassilopoulos D, Tousoulis D, De Luca G, Giustetto C, Rinaldi M, Oh JK, Klein AL, Brucato A, Adler Y. Anakinra for corticosteroid-dependent and colchicine-resistant pericarditis: The IRAP (International Registry of Anakinra for Pericarditis) study. Eur J Prev Cardiol. 2020 Jun;27(9):956-964. doi: 10.1177/2047487319879534. Epub 2019 Oct 15. PMID 31610707
- [Background] Rasmussen LJH, Petersen JEV, Eugen-Olsen J. Soluble Urokinase Plasminogen Activator Receptor (suPAR) as a Biomarker of Systemic Chronic Inflammation. Front Immunol. 2021 Dec 2;12:780641. doi: 10.3389/fimmu.2021.780641. eCollection 2021. PMID 34925360
- [Background] Hodges GW, Bang CN, Wachtell K, Eugen-Olsen J, Jeppesen JL. suPAR: A New Biomarker for Cardiovascular Disease? Can J Cardiol. 2015 Oct;31(10):1293-302. doi: 10.1016/j.cjca.2015.03.023. Epub 2015 Mar 25. PMID 26118447
- [Background] Velissaris D, Zareifopoulos N, Koniari I, Karamouzos V, Bousis D, Gerakaris A, Platanaki C, Kounis N. Soluble Urokinase Plasminogen Activator Receptor as a Diagnostic and Prognostic Biomarker in Cardiac Disease. J Clin Med Res. 2021 Mar;13(3):133-142. doi: 10.14740/jocmr4459. Epub 2021 Mar 19. PMID 33854652
- [Background] Pisacreta AM, Mascolo R, Nivuori M, Dominioni CC, Gabiati C, Trotta L, Pancrazi M, Marco GD, Carollo C, Pedroli A, Casarin F, Tombetti E, Bizzi E, Imazio M, Brucato A. Acute pericarditis with pleuropulmonary involvement, fever and elevated C-reactive protein: A systemic autoinflammatory disease? A cohort study. Eur J Intern Med. 2023 Jul;113:45-48. doi: 10.1016/j.ejim.2023.03.034. Epub 2023 Apr 15. PMID 37069014